CLINICAL TRIAL: NCT03358641
Title: The Relationship Between Physical Activity and Radiographic Osteoarthritis Worsening: Wuchuan Osteoarthritis Study
Brief Title: The Relationship Between Physical Activity and Radiographic Osteoarthritis Worsening
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Lin Chutong, arthritis clinic and research center, Peking University People's Hospital
Other Study IDs: PKUPHOSM
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis, Knee
Keywords: exercise; physical activity; radiographic osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wuchuan residents: All residents that meet the criteria can be enrolled in this group, receiving a home interview (including IPA-Q to assess the level of physical activity) and a weight-bearing posteroanterior semiflexed view of radiographs at tibiofemoral (TF) joints at baseline and 3 years later.
  Interventions: Other: level of physical activity

INTERVENTIONS:
Other: level of physical activity — According to the result of IPA-Q questionnaire, participants are divided in three groups: low level, moderate level, high level of physical activity.

SUMMARY:
Wuchuan Osteoarthritis Study is a population-based longitudinal study of natural history of knee osteoarthritis and its risk factors. At baseline and follow-up visits, IPA-Q questionnaire and a radiographs at tibiofemoral (TF) joints will be taken in order to assess the relationship between physical activity and radiographic osteoarthritis worsening.

DETAILED DESCRIPTION:
1025 residents aged ≥ 50 years will be recruited using door-to-door enumeration in randomly selected rural communities in Wuchuan, China, and will be followed in 3 years. At baseline and follow-up visits, subjects will complete a home interview (including, but not limited to, socio-demographic factors, physical activity level using IPA-Q questionnaire,WOMAC questionnaire) and have a weight-bearing posteroanterior semiflexed view of radiographs at tibiofemoral (TF) joints. Radiographic osteoarthritis (ROA) worsening for a knee is defined if its Kellgren and Lawrence (K/L) grade increases by at least 1 grade except for the change from 0 to 1 during follow-up. The relationship between level of physical activity and ROA worsening will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. people aged 50 or over
2. Wuchuan permanent resident population

Exclusion Criteria:

1. patients with rheumatoid arthritis
2. the disabled
3. patients with mental disorders
4. laid up for malignant tumor
5. people who live or work outside for more than half a year

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People, over 50 years old, in a rural area in Northern China (Wuchuan, Inner Mongolia)
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
worsening of radiographic osteoarthritis | 3 years after enrollment
  The tibiofemoral radiograph of both knee joint will be taken at baseline and in 3 years. Knee radiographs will be read by one investigator according to Kellgren and Lawrence (K/L) criteria. A knee will be defined as ROA worsening if its K/L grade increased by at least 1 grade except for the change from 0 to 1 during follow-up.

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index | 3 years after enrollment
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be assessed at baseline and in 3 years, from which symptoms of patients can be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, MD, Principal Investigator — arthritis clinic and research center

IPD SHARING:
Plan to Share IPD: No